CLINICAL TRIAL: NCT02670317
Title: Multicenter Phase II Single Arm Open-label Study on the Feasibility, Safety and Efficacy of Combination of CHOP-21 Supplemented With Obinutuzumab and Ibrutinib in Untreated Young High Risk Diffuse Large B-cell Lymphoma (DLBCL) Patients.
Brief Title: Phase II Study About Combination CHOP-21, Obinutuzumab and Ibrutinib in Untreated Young High Risk DLBCL Patients.
Acronym: FIL-GALILEO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: GA101-CHOP not advantage from rituximab-CHOP
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL-GALILEO; 2015-005273-20 (EudraCT Number)
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma, B-Cell
Keywords: DLBCL; large B cell lymphoma; NHL
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — obinutuzumab; ibrutinib; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G CHOP 21 + Ibrutinib (Experimental): Patients will receive a maximum of 6 courses of G-CHOP-21 followed by 2 doses of Obinutuzumab in combination with Ibrutinib.
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib; Drug: CHOP

INTERVENTIONS:
Drug: Obinutuzumab — Patients will receive a maximum of 6 courses of G-CHOP-21 followed by 2 doses of Obinutuzumab in combination with Ibrutinib.
  Other Names: GA101
Drug: Ibrutinib — Patients will receive a maximum of 6 courses of G-CHOP-21 followed by 2 doses of Obinutuzumab in combination with Ibrutinib.
  Other Names: Imbruvica
Drug: CHOP — Patients will receive a maximum of 6 courses of CHOP-21 in combination with Obinutuzumab (G) followed by 2 doses of Obinutuzumab in combination with Ibrutinib.
  Other Names: Cyclophosphamide, doxorubicin, vincristine, and prednisone; Hydroxydaunomycin, Oncovin

SUMMARY:
This is a prospective, multicenter, single arm, phase II trial in young patients (18-60 years) with poor-prognosis (aaIPI 2 or 3) newly diagnosed Diffuse Large B-cell Lymphoma (DLBCL).

Aim of the study is to assess the efficacy and the safety of G-CHOP in combination with ibrutinib.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, phase II trial in young patients (18-60 years) with poor-prognosis (age-adjusted International Prognostic Index, aaIPI, 2 or 3) newly diagnosed Diffuse Large B-cell Lymphoma (DLBCL).

Patient will receive 6 courses of G-CHOP21 (Obimutizumab- cyclophosphamide, hydroxydaunomycin, Oncovin, and prednisone) followed by 2 doses of Obinutuzumab supplemented with Ibrutinib. Duration of treatment will be 5 months plus 4-5 weeks for response evaluation.

During the study, disease status will be evaluated after the 4th cycle by computed tomography (CT) scan, and after end of treatment by imaging test (18FDG-PET [positron emission tomography] and CT scan).

Patients will be recruited over 2 years and followed for a minimum of 2 years after the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Diffuse Large B-Cell Lymphoma (DLBCL) not otherwise specified (NOS)
* Previously untreated disease
* Age 18-60
* Age adjusted IPI=2-3
* Ann Arbor stage II-IV disease
* Measurable disease ≥ 1.5 cm in longest diameter, and measurable in 2 perpendicular dimensions
* Normal blood count as defined as: absolute neutrophil count ≥1.0 × 109/L independent of growth factor support, platelet count ≥ 100,000/mm3 or ≥50,000/mm3 if bone marrow (BM) involvement independent of transfusion support in either situation
* Normal organ functions defined as: creatinine ≤2 times the upper limit of normal (ULN) or estimated Glomerular Filtration Rate (Cockroft- Gault) ≥40 ml/min/1.73m2, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3× the ULN; total bilirubin ≤ 1.5 × the ULN unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN; International normalized ratio (INR) < 1.5 × the ULN in the absence of therapeutic anticoagulation; partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) < 1.5 × the ULN in the absence of a lupus anticoagulant"
* Patients with occult or prior hepatitis B infection (defined as HBsAg negative, anti-HBs positive and /or anti-HBc positive) may be included if hepatitis B virus (HBV) DNA is undetectable. These patients must be willing to undergo bi-monthly DNA testing and they should receive prophylaxis with Lamivudine
* No active hepatitis C virus (HCV) infection
* Known availability of biopsy material
* No Central Nervous System (CNS) disease (meningeal and/or brain involvement by lymphoma)
* Absence of active infections
* Non peripheral neuropathy or active neurological non neoplastic disease of CNS
* Non major surgical intervention prior 3 months to enrolment if not due to lymphoma and/or not other disease life-threatening that can compromise chemotherapy treatment
* Patient with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study.
* Patients with any other malignancy that has been treated with surgery alone with curative intent and the malignancy has been in remission without treatment for at least 5 years prior to enrolment.
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 6 months after the last dose of study drug. For males, these restrictions apply for 6 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (betahuman chorionic gonadotropin [β-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Life expectancy > 6 months
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Any Other histologies than Diffuse Large B- Cell Lymphoma (DLBCL): composite or transformed disease and patients with follicular lymphoma IIIB
* Primary mediastinal lymphoma (PMBL)
* Known central nervous system lymphoma
* Any prior lymphoma therapy
* Contraindication to any drug in the chemotherapy regimen
* Left ventricular ejection fraction (LVEF) < 50%
* Neuropathy ≥ grade 2
* Seropositive for or active viral infection with HBV
* HBsAg positive
* HBsAg negative, anti-HBs positive and /or anti-HBc positive with detectable viral DNA
* Known seropositive active HCV
* Human immunodeficiency virus (HIV) infection
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma): creatinine ≥ 2 times the ULN (unless creatinine clearance normal, or calculated creatinine clearance < 40 mL/min (using the Cockcroft-Gault formula); AST or ALT ≥3 × the ULN; total bilirubin >1.5 × the ULN: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN; INR > 1.5 × the ULN in the absence of therapeutic anticoagulation; PTT or aPTT > 1.5 × the ULN in the absence of a lupus anticoagulant"
* History of stroke or intracranial hemorrhage within the past 6 months.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Presence of major neurological disorders
* any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
* Major surgical intervention prior 4 weeks to enrollment if not due to lymphoma and/or other disease life-threatening that can compromise chemotherapy treatment
* Prior malignancies other than lymphoma in the last 5 years with exception of currently treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix
* Any other coexisting medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
* If female, the patient is pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The efficacy of G-CHOP-21 in combination with Ibrutinib in terms of 2-yrs PFS (progression-free survival) | 2 years
The safety of G-CHOP-21 in combination with Ibrutinib in terms of proportion of patients experiencing grade 3 or greater extra-hematologic toxicity or treatment interruption for safety reasons or any toxic death during the 6 cycles of treatment | 5 months of treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
Complete Remission (CR) Rate | 6 months
Overall Response Rate (ORR) | 6 months
The Duration Of Response (DOR) after the end of treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Martelli, MD, Principal Investigator — Policlinico Umberto I - Università "La Sapienza"
Locations (29):
- Italy (29):
  - IRCCS Candiolo - Fondazione del Piemonte per l'oncologia, Candiolo, TO
  - AO SS. Antonio e Biagio e C. Arrigo, Alessandria
  - AOU Policlinico Consorziale, Bari
  - AO Papa Giovanni XXIII, Bergamo
  - Ospedale di Bolzano, Bolzano
  - Ospedale Businco, Cagliari
  - AO di Cosenza, Cosenza
  - AOU Careggi, Florence
  - P.O. Vito Fazzi, Lecce
  - IRST Meldola, Meldola
  - Ospedale Papardo, Messina
  - Istituto Europeo Oncologico, Milan
  - AOU Policlinico di Modena, Modena
  - Ospedale San Gerardo, Monza
  - IRCCS Napoli Pascale, Napoli
  - Ospedale Maggiore della Carità, Novara
  - AOOR Villa Sofia Cervello, Palermo
  - AOU di Parma, Parma
  - Ospedale G. Da Saliceto, Piacenza
  - AOR San Carlo, Potenza
  - Ospedale Degli Infermi, Rimini
  - Policlinico Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Humanitas, Rozzano
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - AOU Città Della Salute e Della Scienza Ematologia Universitaria, Torino
  - AOU Città Della Salute e Della Scienza SC Ematologia, Torino
  - AOU di Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: No